CLINICAL TRIAL: NCT02933762
Title: An Exploratory, Single-Blind, Placebo-Controlled, Randomized, Single- and Multiple-Dose Pharmacodynamics Study in Healthy Subjects to Evaluate the Effect of JNJ-54175446 on Amyloid Biomarkers and Cytokine Profiles in Cerebrospinal Fluid and Plasma
Brief Title: A Study in Healthy Participants to Evaluate the Effect of JNJ-54175446 on Amyloid Biomarkers and Cytokine Profiles in Cerebrospinal Fluid and Plasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR108231; 2016-003040-37 (EudraCT Number); 54175446EDI1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-09-21; First posted 2016-10-14 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-54175446

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (13):
- Part 1: Cohort A1 (JNJ-54175446 30 milligram[mg]) (Experimental): Healthy elderly participants will receive single dose of 30mg JNJ-54175446.
  Interventions: Drug: JNJ-54175446
- Part 1: Cohort A1 (JNJ-54175446 100mg) (Experimental): Healthy elderly participants will receive single dose of 100mg JNJ-54175446.
  Interventions: Drug: JNJ-54175446
- Part 1: Cohort A1 (JNJ-54175446 300mg) (Experimental): Healthy elderly participants will receive single dose of 300mg JNJ-54175446.
  Interventions: Drug: JNJ-54175446
- Part 1: Cohort A1 (Placebo) (Experimental): Healthy elderly participants will receive single dose of placebo.
  Interventions: Drug: Placebo
- Part 1: Cohort A2 (JNJ-54175446 D1 mg) (Experimental): Healthy elderly participants will receive an additional dose D1 mg [less than or equal to (<=) 600 mg] of JNJ-54175446, to be determined.
  Interventions: Drug: JNJ-54175446
- Part 1: Cohort A3 (JNJ-54175446 D2 mg) (Experimental): Healthy young participants will receive a single dose D2 mg (<= 600 mg) of JNJ-54175446, to be determined.
  Interventions: Drug: JNJ-54175446
- Part 1: Cohort A3 (Placebo) (Experimental): Healthy young participants will receive a single dose of placebo.
  Interventions: Drug: Placebo
- Part 2: Cohort B1 (JNJ-54175446 D3 mg) (Experimental): Healthy elderly participants will receive multiple dose levels D3 mg (<= 450 mg) of JNJ-54175446 determined based on the results from Cohort A1.
  Interventions: Drug: JNJ-54175446
- Part 2: Cohort B1 (Placebo) (Experimental): Healthy elderly participants will receive placebo determined based on the results from Cohort A1.
  Interventions: Drug: Placebo
- Part 2: Cohort B2 (JNJ-54175446 D4 mg) (Experimental): Healthy elderly participants will receive multiple dose levels D4 mg (<= 450 mg) of JNJ-54175446 determined based on the results from Cohort A1.
  Interventions: Drug: JNJ-54175446
- Part 2: Cohort B2 (Placebo) (Experimental): Healthy elderly participants will receive placebo determined based on the results from Cohort A1
  Interventions: Drug: Placebo
- Part 2: Cohort B3 (JNJ-54175446 D5 mg) (Experimental): Healthy elderly participants will receive multiple dose levels D5 mg (<= 450 mg) of JNJ-54175446 determined based on the results from Cohort A1.
  Interventions: Drug: JNJ-54175446
- Part 2: Cohort B3 (Placebo) (Experimental): Healthy elderly participants will receive placebo determined based on the results from Cohort A1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54175446 — Participants will receive a single oral dose of JNJ-54175446 suspension orally once on Day 1 of part 1 and Day 1 to Day 7 in part 2.
  Arms: Part 1: Cohort A1 (JNJ-54175446 100mg); Part 1: Cohort A1 (JNJ-54175446 30 milligram[mg]); Part 1: Cohort A1 (JNJ-54175446 300mg); Part 1: Cohort A2 (JNJ-54175446 D1 mg); Part 1: Cohort A3 (JNJ-54175446 D2 mg); Part 2: Cohort B1 (JNJ-54175446 D3 mg); Part 2: Cohort B2 (JNJ-54175446 D4 mg); Part 2: Cohort B3 (JNJ-54175446 D5 mg)
Drug: Placebo — Participants will receive a single oral dose of JNJ-54175446 suspension orally once on Day 1 of part 1 and Day 1 to Day 7 in part 2.
  Arms: Part 1: Cohort A1 (Placebo); Part 1: Cohort A3 (Placebo); Part 2: Cohort B1 (Placebo); Part 2: Cohort B2 (Placebo); Part 2: Cohort B3 (Placebo)

SUMMARY:
The primary purpose of this study is to investigate the effects of JNJ-54175446 (dose response) on levels of Aβ fragments (Aβ1-42, Aβ1-40, Aβ1-38, Aβ1-37) in plasma and cerebrospinal fluid (CSF), the effects of JNJ-54175446 on markers of (neuro) inflammation/protection in blood and CSF and the pharmacokinetics of JNJ-54175446 followed by single and multiple dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) between 18 and 32 kilogram (kg)/ meter (m)^2, inclusive (BMI = weight/height^2)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG)

Part 1 and 2 (Elderly Participants):

* Healthy male or female participants between 55 and 75 years of age, inclusive
* Participant must be healthy on the basis of both physical and neurological examination performed at Screening and at admission to the clinical unit

Part 1 (Young Participants):

- Healthy male participants between 18 and 45 years of age, inclusive

Exclusion Criteria:

* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the participant
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening (per Screening evaluations)
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening (per Screening evaluations)
* Participant has a history of malignancy within 5 years before Screening
* Participant has signs of increased intracranial pressure based on fundoscopy at Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The Effects of JNJ-54175446 (Dose Response) on Levels of Aβ Fragments in Plasma | Part 1: Up to Day 2
The Effects of JNJ-54175446 (Dose Response) on Levels of Aβ Fragments in Plasma | Part 2: Up to Day 8
The Effects of JNJ-54175446 (Dose Response) on Levels of Aβ Fragments in Cerebrospinal Fluid (CSF) | Part 1: Up to Day 2
The Effects of JNJ-54175446 (Dose Response) on Levels of Aβ Fragments in Cerebrospinal Fluid (CSF) | Part 2: Up to Day 8
The Effects of JNJ-54175446 (Dose Response) on Markers of (Neuro)Inflammation / Protection in Blood | Part 1: Up to Day 2
The Effects of JNJ-54175446 (Dose Response) on Markers of (Neuro)Inflammation / Protection in Blood | Part 2: Up to Day 8
The Effects of JNJ-54175446 (Dose Response) on Markers of (Neuro)Inflammation / Protection in CSF | Part 1: Up to Day 2
The Effects of JNJ-54175446 (Dose Response) on Markers of (Neuro)Inflammation / Protection in CSF | Part 2: Up to Day 8
Maximum Observed Plasma Concentration (Cmax) After Single- and Multiple-Dose Administration | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
Minimum Observed Plasma Concentration (Cmin)During Dosing Interval | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
The Observed Plasma Concentration Just Prior to the Beginning or at the end of a Dosing Interval of any Dose Other Than the First Dose (Ctrough) | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
Average Plasma Concentration at Steady State Over the Dosing Interval (Cavg) | Part 1: Day 1 - Day 2; Par 2: Day 1, Day 2 to 6, Day 7, Day 8
Time to Reach the Maximum Plasma Concentration, After Single- and Multiple-Dose Administration (Tmax) | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
Area Under The Concentration-Time Curve From 0 To t Hours Postdosing (AUCt) | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
Area Under the Concentration-Time Curve From 0 to 24 Hours Postdosing (AUC24h) | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8
The Ratio of the Maximum Plasma Concentration (Peak) to Trough Observed Concentration (Peak/Trough Ratio) | Part 1: Day 1 - Day 2; Part 2: Day 1 to Day 8

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Screening up to follow-up (in part 1 and part 2 [approximately up to 8 weeks])

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Triana-Baltzer G, Timmers M, De Boer P, Schoene M, Furey M, Bleys C, Vrancken I, Slemmon R, Ceusters M, van Nueten L, Kolb H. Profiling classical neuropsychiatric biomarkers across biological fluids and following continuous lumbar puncture: A guide to sample type and time. Compr Psychoneuroendocrinol. 2022 Jan 15;10:100116. doi: 10.1016/j.cpnec.2022.100116. eCollection 2022 May. PMID 35774109